CLINICAL TRIAL: NCT03167164
Title: NANT Merkel Cell Carcinoma (MCC) Vaccine: Combination Immunotherapy in Subjects With MCC Who Have Progressed on or After Anti-programmed Death-ligand 1 (PD-L1) Therapy
Brief Title: QUILT-3.045: NANT Merkel Cell Carcinoma (MCC) Vaccine: Combination Immunotherapy in Subjects With MCC Who Have Progressed on or After PD-L1 Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.045
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2017-10

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab; Bevacizumab; Capecitabine; Cisplatin; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Omacor; Radiosurgery; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT MCC Vaccine (Experimental): A combination of agents will be administered to subjects in this study:
  avelumab, bevacizumab, capecitabine, cisplatin, cyclophosphamide, 5-fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ethyl esters, stereotactic body radiation therapy, ALT-803, ETBX-051, ETBX-061, GI-6301, and haNK.
  Interventions: Biological: Avelumab; Biological: Bevacizumab; Drug: Capecitabine; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: 5-fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: omega-3-acid ethyl esters; Radiation: Stereotactic Body Radiation Therapy; Biological: ALT-803; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-6301; Biological: haNK

INTERVENTIONS:
Biological: Avelumab — Fully human anti-PD-L1 IgG1 lambda monoclonal antibody
Biological: Bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal antibody
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cisplatin — (SP-4-2)-diamminedichloroplatinum(II)
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: 5-fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — Calcium N-[p-[[[(6RS)-2-amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl]methyl]amino]benzoyl]-L-glutamate (1:1)
Drug: nab-Paclitaxel — 5β,20-Epoxy-1,2α,4,7β,10β,13α-hexahydroxytax-11-en-9-one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)-N-benzoyl-3-phenylisoserine
Drug: omega-3-acid ethyl esters — Omega-3-acid ethyl esters
Radiation: Stereotactic Body Radiation Therapy — radiation
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury
Biological: ETBX-061 — Ad5 [E1-, E2b-]-MUC1
Biological: GI-6301 — Heat-killed S. cerevisiae yeast expressing the human Brachyury (hBrachyury) oncoprotein
Biological: haNK — NK-92 [CD16.158V, ER IL-2] (high-affinity activated Natural Killer cells)

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with MCC who have progressed on or after anti-PD-L1 therapy.

DETAILED DESCRIPTION:
Treatment will be administered in two phases. Subjects will continue treatment until they experience progressive disease (PD) or experience unacceptable toxicity (not correctable with dose reduction), withdraw consent, or if the investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) will enter phase 2 of the study. Subjects may remain on phase 2 of the study for up to 1 year. Treatment will continue in phase 2 until the subject experiences PD or unacceptable toxicity (not correctable with dose reduction), withdraws consent, or if the investigator feels it is no longer in the subject's best interest to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed metastatic or unresectable MCC with progression on or after anti-PD-L1 therapy (eg, avelumab).
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.5 cm.
6. Must have a recent tumor biopsy specimen obtained following the conclusion of the most recent anti-cancer treatment. If a historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period.
7. Must be willing to provide blood samples for exploratory analyses, and if considered safe by the investigator, a tumor biopsy specimen at 8 weeks after the start of treatment.
8. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment.

Exclusion Criteria:

1. History of persistent grade 2 or higher (CTCAE Version 4.03) hematologic toxicity resulting from previous therapy.
2. History of other active malignancies or brain metastasis except: controlled basal cell carcinoma; prior history of in situ cancer (eg, breast, melanoma, cervical); prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy) and with undetectable PSA (< 0.2 ng/mL); bulky (≥ 1.5 cm) disease with metastasis in the central hilar area of the chest and involving the pulmonary vasculature. Subjects with a history of another malignancy must have > 5 years without evidence of disease.
3. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
4. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
5. History of organ transplant requiring immunosuppression.
6. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
7. Requires whole blood transfusion to meet eligibility criteria.
8. Inadequate organ function, evidenced by the following laboratory results:

   1. WBC count < 3,500 cells/mm3.
   2. Absolute neutrophil count < 1,500 cells/mm3.
   3. Platelet count < 100,000 cells/mm3.
   4. Hemoglobin < 9 g/dL.
   5. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   6. AST (SGOT)) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   7. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   8. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   9. INR or aPTT or PTT >1.5 × ULN (unless on therapeutic anti-coagulation).
9. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
10. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
11. Positive results of screening test for HIV, HBV, or HCV.
12. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
13. Known hypersensitivity to any component of the study medication(s).
14. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
15. Concurrent or prior use of a strong CYP3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
16. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
17. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
18. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
19. Concurrent participation in any interventional clinical trial.
20. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), graded using the NCI CTCAE Version 4.03. | 1 year
  Phase 1b primary endpoint
Objective response rate by RECIST Version 1.1 | 1 year
  Phase 2 primary endpoint
Objective response rate by irRC | 1 year
  Phase 2 primary endpoint

SECONDARY OUTCOMES:
Objective response rate by RECIST Version 1.1 | 1 year
  Phase 1b secondary endpoint
Objective response rate by irRC | 1 year
  Phase 1b secondary endpoint
Progression-free survival by RECIST Version 1.1 | 2 years
  Phase 1b and Phase 2 secondary endpoint
Progression-free survival by irRC | 2 years
  Phase 1b and Phase 2 secondary endpoint
Overall survival | 2 years
  Phase 1b and Phase 2 secondary endpoint
Duration of response | 2 years
  Phase 1b and Phase 2 secondary endpoint
Disease control rate (confirmed complete response, partial response, or stable disease lasting for at least 2 months) | 2 years
  Phase 1b and Phase 2 secondary endpoint
Quality of life by patient-reported outcome using Functional Assessment of Cancer Therapy-Melanoma (FACT-M) Questionnaire | 2 years
  Phase 1b and Phase 2 secondary endpoint
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), graded using the NCI CTCAE Version 4.03 | 1 year
  Phase 2 secondary endpoint

IPD SHARING:
Plan to Share IPD: No